CLINICAL TRIAL: NCT02327624
Title: Study of Two Regimens of TicagrElor Compared to Clopidogrel in Patients Undergoing ELective Percutaneous Coronary Intervention
Brief Title: STEEL Percutaneous Coronary Intervention
Acronym: STEEL-PCI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STH18423
Record Dates: First submitted 2014-12-10; First posted 2014-12-30 (Estimated); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Clopidogrel (Active Comparator): The standard antiplatelet treatment for patients is pretreatment with aspirin and clopidogrel. In this trial patients will be randomised in clopidogrel orTicagrelor of two doses
  Interventions: Drug: Clopidogrel
- Ticagrelor 60 (Experimental): Ticagrelor 60 is a new dosage to be tried in this trial.
  Interventions: Drug: Ticagrelor 60
- Ticagrelor 90 (Experimental): Ticagrelor 90 is used following clopidogrel as maintenance therapy with aspirin 75 mg daily and clopidogrel 75 mg daily following PCI for at least 1 month.
  Interventions: Drug: Ticagrelor 90

INTERVENTIONS:
Drug: Clopidogrel — Compare Clopidogrel to two doses of Ticagrelor 60 and 90
  Arms: Clopidogrel
Drug: Ticagrelor 60 — Compare Clopidogrel to two doses of Ticagrelor 60 and 90
  Arms: Ticagrelor 60
Drug: Ticagrelor 90 — Compare Clopidogrel to two doses of Ticagrelor 60 and 90
  Arms: Ticagrelor 90

SUMMARY:
The principal hypothesis of this study is that two different maintenance regimens of ticagrelor are safe, tolerable and associated with significant inhibition of erythrocyte adenosine reuptake compared to clopidogrel in patients undergoing elective Percutaneous Coronary Intervention (PCI) for stable Coronary artery disease (CAD).

DETAILED DESCRIPTION:
Coronary artery disease (CAD) is caused by fatty deposits building up over time in the arteries that supply the heart with blood, causing the arteries to narrow and reducing the amount of blood that can get to the heart. One of the treatment options for CAD is percutaneous coronary intervention (PCI) in which a balloon is inserted into the artery supplying the heart to open up the artery where it has narrowed. A stent is then left in the artery once the balloon is removed to hold the artery open and allow more blood to flow to the heart. One of the risks of this procedure, as in CAD itself, is the formation of blood clots that then block the arteries, stopping or reducing blood flow and causing a heart attack.

Platelets are small blood cells involved in the formation of blood clots that cause heart attacks. Antiplatelet drugs (e.g. aspirin) are given to patients with CAD to reduce the risk of a clot forming in the future and causing a heart attack. In a recent large clinical trial (PLATO study), it was shown that heart attack patients treated with a new antiplatelet medication (ticagrelor) had fewer later heart attacks compared to the current standard treatment (clopidogrel). The STEELPCI study is comparing three different strategies for prescribing antiplatelet medication to patients with stable CAD who have a PCI.

Patients on waiting list for PCI who meet the study inclusion/exclusion criteria will be invited to participate. Patients will have their PCI as normal but be randomised to take one of three different medication strategies, either clopidogrel or one of two doses of ticagrelor. Patient will take the medication for 30 days and have blood tests and meet with the research team during that time to assess the effects of each medication strategy.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent prior to any study specific procedures
2. Male or female aged greater than 18 years
3. Previous invasive coronary angiography with plan for PCI with coronary stent implantation for stable coronary artery disease

Exclusion Criteria:

1. Requirement for a chronic total occlusion to be crossed in order for any stent implantation to proceed
2. Plan for coronary angiography with a view to PCI if appropriate (i.e. current coronary anatomy not known)
3. Intention to use platelet function tests or genotyping to guide antiplatelet therapy
4. Known allergy to or intolerance of aspirin, clopidogrel or ticagrelor
5. Treatment with antiplatelet medication apart from aspirin or clopidogrel that cannot be stopped 10 days prior to PCI (e.g. ticagrelor, prasugrel, dipyridamole, ticlopidine, abciximab, tirofiban), for example because of continuing indication
6. Planned treatment or consideration of treatment with oral antiplatelet medication other than aspirin or clopidogrel following PCI
7. Planned use of a glycoprotein IIb/IIIa antagonist for the PCI procedure
8. Myocardial infarction within the past 12 months
9. Current or planned use of an oral anticoagulant (e.g. warfarin, dabigatran, rivaroxaban, apixaban)
10. Previous history of intracranial haemorrhage or other intracranial pathology associated with increased bleeding risk
11. Haemoglobin < 100 g/L or other evidence of active bleeding
12. Peptic ulceration documented by endoscopy within the last 3 months unless healing proven by repeat endoscopy
13. History of acute or chronic liver disease (e.g. cirrhosis)
14. Treatment in the last 10 days or requirement for ongoing treatment with a strong CYP3A4 inhibitor or inducer (see section 5.6.8)
15. Requirement for ongoing treatment with simvastatin or lovastatin at a dose greater than 40 mg per day
16. Treatment with a CYP3A4 substrate with a narrow therapeutic index (e.g. cyclosporine, quinidine)
17. End-stage renal failure requiring dialysis
18. History of alcohol or drug abuse in the last year
19. Co-morbidity associated with life expectancy less than 1 year
20. Females of child-bearing potential unless negative pregnancy test at screening and willing to use effective contraception (i.e. established use of oral, injected or implanted hormonal methods of contraception or placement of an intrauterine device (IUD) or intrauterine system (IUS) or barrier methods of contraception with spermicide or sole male partner with prior vasectomy and confirmed absence of sperm in ejaculate) for the duration of treatment with study medication
21. Any other condition deemed by the investigator to place the patient at excessive risk of bleeding with ticagrelor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
Platelet function in the three treatment groups | 2 years

SECONDARY OUTCOMES:
Rates of myocardial infarction following PCI | 2 years
Plasma adenosine concentration in the three treatment groups | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Sheffield Teaching Hospitals NHS FT, Sheffield, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Orme RC, Parker WAE, Thomas MR, Judge HM, Baster K, Sumaya W, Morgan KP, McMellon HC, Richardson JD, Grech ED, Wheeldon NM, Hall IR, Iqbal J, Barmby D, Gunn JP, Storey RF. Study of Two Dose Regimens of Ticagrelor Compared With Clopidogrel in Patients Undergoing Percutaneous Coronary Intervention for Stable Coronary Artery Disease. Circulation. 2018 Sep 25;138(13):1290-1300. doi: 10.1161/CIRCULATIONAHA.118.034790. Epub 2018 Jul 24. PMID 29930021